CLINICAL TRIAL: NCT02844283
Title: Adenovirus Carrying Hepatocyte Growth Factor (Ad-HGF) Treatment for Myocardial Infarction
Brief Title: Ad-HGF Treatment for Myocardial Infarction
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-6-29
Record Dates: First submitted 2016-06-29; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-06

CONDITIONS: Myocardial Infarction
Keywords: HGF,myocardial infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- treatment group (Experimental): Single dose of Ad-HGF given by investigator via intracoronary injection into infarct-related artery
  Interventions: Drug: Ad-HGF
- control group (Sham Comparator): 0.9% sodium chloride (NaCl) injection of same volume given by investigator via intracoronary injection into infarct-related artery
  Interventions: Other: 0.9% NaCl

INTERVENTIONS:
Drug: Ad-HGF
  Arms: treatment group
Other: 0.9% NaCl
  Arms: control group

SUMMARY:
This will be the first clinical trial use Ad-HGF gene for the treatment of myocardial infarction disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-80 years of age

  * Clinical diagnosis of anterior ST-segment elevation myocardial infarction (STEMI) within the last 30 days, with any one of the following 12-lead electrocardiographic changes:
  * a) Greater than or equal to 2 mm ST-segment elevation) in 2 adjacent electrocardiographic precordial leads
  * b) A new left bundle branch block AND and an increase in cardiospecific enzymes >3x CK, or increase in troponin compared to institution laboratory normal ranges
  * Successful PCI with stent implantation to infarct-related artery within the last 30 days; defined as residual stenosis no greater than 30%, Thrombolysis In Myocardial Infarction (TIMI) flow of at least 2 and a reference diameter of at least > 2mm
  * Is considered hemodynamically stable at time of enrollment and immediately prior to Ad-HGF delivery
  * Screening LVEF for the first 12 enrolled participants, must be no greater than 40% by echocardiography (determined by Simpson's method) performed at least 2 days after revascularization procedure. Subsequent participants enrolled in the trial, must have an LVEF no greater than 45%. (All screening echos done within the first 4 days post percutaneous coronary intervention (PCI) must be repeated either by echocardiography or MRI prior to Ad-HGF delivery to ensure that the variability does not exceed 10%)
  * In the case of a previous myocardial infarction, documented LVEF must be 50% or greater
  * Female participants must be surgically sterile, post-menopausal, have documented infertility, or are of child-bearing potential wih laboratory confirmation of non-pregnant state
  * Provided written informed consent and is willing to comply with study follow-up visits

Exclusion Criteria:

* Significant unprotected left main disease (stenosis of 50% or greater)on diagnostic angiography

  * An increase in LVEF by greater that 10% from initial LVEF evaluation for repeat assessments
  * The presence of significant coronary lesions, other than the index lesion of the infarction related artery
  * A history of significant ventricular arrhythmia not related to index STEMI
  * A history of cerebro-vascular accident or transient ischemic attack within 6 months of enrollment
  * Inability to undergo apheresis procedure(i.e.: poor venous access, laboratory abnormalities
  * A history of uncorrected significant valvular heart disease
  * A history of left ventricular dysfunction prior to index STEMI
  * A history of human immunodeficiency virus (HIV)or hepatitis B or C infection
  * A history of malignancy within 5 years (Except for low-grade and fully resolved non-melanoma skin cancer)
  * A history of allergy to gentamycin or amphotericin
  * A history of non-compliance
  * Active inflammatory autoimmune disease requiring chronic immunosuppressive therapy
  * Creatinine clearance <60 by Cockcroft-Gault Calculator
  * Confirmed pregnant or lactating
  * Is enrolled in a current investigational drug or device trial
  * Participant has received cell or gene therapy in past
  * The presence of any significant co-morbidities that, in the investigator's opinion, would preclude the participant from taking part in the trial
  * Inability to provide informed consent and comply with the follow-up visit schedule

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
changes of cardiac left ventricular ejection fraction (LVEF, %) | Baseline to 6 months
  the difference of LVEF before and after treatment between groups.

SECONDARY OUTCOMES:
Quality of Life Measures (SF-36) | Baseline to 6 months
  Participants will complete SF-36 to measure quality of life at baseline, 3 and 6 months.
Activity Status (DASI) | Baseline to 6 months
  Participants will complete DASI questionnaires to measure activity status at baseline, 3 and 6 months.
changes of creatinine kinase (CK, U/L) within 24 hours post delivery. | Baseline to 24 hours post delivery.
  the difference of creatinine kinase (CK, U/L) before and after delivery within 24 hours.
changes of troponin (μg/L) within 24 hours post delivery. | Baseline to 24 hours post delivery.
  the difference of troponin (μg/L) before and after delivery within 24 hours
number of participants with evidence of any systemic embolization within 1 week post delivery. | Baseline to 1 week post delivery.
  number of participants with evidence of any systemic embolization during the hospitalization period post delivery.
number of participants with clinically significant changes in ECG than before | Baseline to 6 months
  number of participants with clinically significant changes in ECG than before
number of participants with major acute cardiac events (cardiac death and myocardial infarction) during follow-up | Baseline to 6 months
  number of participants with major acute cardiac events (cardiac death and myocardial infarction) during follow-up
number of participants with revascularization procedures during follow-up | Baseline to 6 months
  number of participants with revascularization procedures during follow-up